CLINICAL TRIAL: NCT00721968
Title: A Prospective, Randomized, Controlled, Parallel Groups, Multicenter Clinical Investigation Of The Trabecular Micro-Bypass Stent Model GTS400 In Conjunction With Cataract Surgery
Brief Title: Safety and Efficacy of the GTS400 Stent in Conjunction With Cataract
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Glaukos Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GC-005
Record Dates: First submitted 2008-07-23; First posted 2008-07-25 (Estimated); Results first posted 2014-03-06 (Estimated); Last update posted 2014-03-06 (Estimated); Status verified 2014-02

CONDITIONS: Open-angle Glaucoma
Keywords: Open angle; Glaucoma; Cataract; Surgery
MeSH Terms: conditions — Glaucoma, Open-Angle; Glaucoma; Cataract | interventions — Cataract Extraction; Phacoemulsification

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Treatment Group (Group 1): Glaukos Trabecular Micro-Bypass Stent Model GTS400; implantation in conjunction with cataract surgery
  Interventions: Device: Glaucoma Stent Surgery (GTS400 Stent)
- 2 (Placebo Comparator): Control Group (Group 2): Cataract surgery only
  Interventions: Procedure: cataract surgery alone

INTERVENTIONS:
Device: Glaucoma Stent Surgery (GTS400 Stent) — ab interno trabecular bypass stent surgery
  Other Names: GTS400 Stent
  Arms: 1
Procedure: cataract surgery alone — Cataract surgery alone
  Other Names: Phacoemulsification
  Arms: 2

SUMMARY:
To evaluate the safety and efficacy of the Glaukos Trabecular Micro-Bypass Stent Model GTS400 in conjunction with cataract surgery, compared to cataract surgery only, in subjects with mild to moderate open angle glaucoma.

DETAILED DESCRIPTION:
The objective of this trial is to evaluate the safety and efficacy of the Glaukos Trabecular Micro-Bypass Stent Model GTS400 (hereinafter referred to as GTS400) in combination with cataract surgery, compared to cataract surgery only, in subjects with mild to moderate primary open-angle glaucoma. This is a prospective, randomized, concurrently controlled, parallel groups, multicenter clinical investigation of the GTS400. Treatment will consist of either implantation of GTS400 stents in the study eye in conjunction with cataract surgery (Group 1, Investigational Group), or cataract surgery only (Group 2, Control Group). Clinical data through 12 months postoperative will form the basis of a pre-market approval (PMA) submission. Subjects will be followed for two years postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Mild to moderate Open-Angle Glaucoma with specific criteria, in need of cataract surgery
* Subject willing to attend scheduled follow-up exams for two years postoperatively, Subject willing to provide written informed consent on the Institutional Review Board approved Informed Consent Form

Exclusion Criteria:

Not meeting inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2007-03; Primary Completion 2012-02 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Head of Clinical Affairs, Study Director — Glaukos Corporation

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 62 enrolled and 44 randomized. Therefore 18 subjects enrolled who either did not pass baseline visit or were not randomized to the trial.
Groups:
- 1 Treatment Group: iStent + Cataract Surgery: Treatment Group (Group 1): Glaukos Trabecular Micro-Bypass Stent Model GTS400; implantation in conjunction with cataract surgery
- 2 Control Group: Cataract Surgery Only: Control Group (Group 2): Cataract surgery only
Period: Overall Study
Arm/Group | 1 Treatment Group: iStent + Cataract Surgery | 2 Control Group: Cataract Surgery Only
Started | 27 | 17
Completed | 25 | 17
Not Completed | 2 | 0
Not completed — Lost to Follow-up | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1 Treatment Group: iStent + Cataract Surgery | 2 Control Group: Cataract Surgery Only | Total
Number analyzed (Participants) | 27 | 17 | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 3 | 4
  >=65 years | 26 | 14 | 40
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 10 | 30
  Male | 7 | 7 | 14
Region of Enrollment [Number; unit: participants]
  United States | 27 | 17 | 44

OUTCOME MEASURES:

1. Primary Outcome: Month 12 Intraocular Pressure ≤ 18 mmHg Without Topical Hypotensive Medications
Description: Percent reaching this endpoint
Time Frame: 12 months
Population: Number of subjects at Month 12 with IOP ≤ 18 mmHg without topical hypotensive medications
Measure: Number; unit: participants
Arm/Group | 1 Treatment Group: iStent + Cataract Surgery | 2 Control Group: Cataract Surgery Only
Number analyzed (Participants) | 27 | 17
participants | 18 | 4

2. Other Pre Specified Outcome: Number of Ocular Hypotensive Medications by Visit
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: medications
Arm/Group | 1 Treatment Group: iStent + Cataract Surgery | 2 Control Group: Cataract Surgery Only
Number analyzed (Participants) | 25 | 17
medications | 0.4 (0.8) | 0.9 (0.7)

ADVERSE EVENTS:
Arm/Group | 1 Treatment Group: iStent + Cataract Surgery | 2 Control Group: Cataract Surgery Only
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/17
Other Adverse Events (participants affected / at risk) | 15/27 | 12/17
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1 Treatment Group: iStent + Cataract Surgery (N=27) | 2 Control Group: Cataract Surgery Only (N=17)
IOP increase >=10 mmHg versus baseline IOP at any visit (Eye disorders) | 3 (3) | 9 (9)
Posterior Capsule Opacification (Eye disorders) | 4 (4) | 1 (1)
Corneal Abrasion (Eye disorders) | 2 (2) | 1 (1)
Conjunctivitis (Eye disorders) | 3 (3) | 2 (2)
Iritis (Eye disorders) | 2 (2) | 0 (0)
Punctate Corneal Staining (Eye disorders) | 1 (1) | 1 (1)
Superficial Punctate Keratitis (Eye disorders) | 1 (1) | 1 (1)
BCVA Loss greater than or equal to 1 line after 3 months post-op (Eye disorders) | 0 (0) | 2 (2)
Eye pain (Eye disorders) | 0 (0) | 2 (2)
Blurry Vision (Eye disorders) | 1 (1) | 1 (1)
Retinal Detachment (Eye disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
There are no limitations and caveats to report

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No